CLINICAL TRIAL: NCT01608763
Title: What is the Active Ingredient in Personalized Feedback Interventions for Problem Drinkers? A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, John Cunningham, Principal Investigator, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 001/2012
Record Dates: First submitted 2012-05-28; First posted 2012-05-31 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Problem Drinking
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Full personalized feedback (Experimental): Participant provided with the full CYD personalized feedback summary.
  Interventions: Behavioral: Check Your Drinking (CYD) personalized feedback intervention
- Only normative feedback (Experimental): Participant provided with just the normative feedback component of the CYD personalized feedback summary.
  Interventions: Behavioral: Check Your Drinking (CYD) personalized feedback intervention
- Just other personalized feedback (Experimental): Participant provided with all the other personalized feedback components of the CYD intervention (i.e., no normative feedback).
  Interventions: Behavioral: Check Your Drinking (CYD) personalized feedback intervention
- No intervention control (No Intervention): Participant provided with a list describing the components of the CYD intervention but not provided any personalized feedback.

INTERVENTIONS:
Behavioral: Check Your Drinking (CYD) personalized feedback intervention — The CYD provides problem drinkers with a personalized summary of their drinking that compares his or her drinking with that of the general population. The CYD also provides an assessment of the severity of the person's drinking problem.
  Arms: Full personalized feedback; Just other personalized feedback; Only normative feedback

SUMMARY:
The major objective of this project is to conduct a randomized controlled trial comparing the impact of the normative feedback and other personalized feedback components of the Check Your Drinking (CYD) Internet-based intervention in the general population. Eligible problem drinking participants will be randomly assigned to one of four conditions in a 2 by 2 design - to receive just the normative feedback component of the CYD intervention, just the other personalized feedback information, to a no intervention control condition, or to receive the full CYD intervention. The no intervention control condition will not be sent any intervention materials but will instead be sent a list of the different components of the CYD feedback and will be asked to think about how useful they would find each of them. All participants will be followed-up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* problem drinkers as measured by an AUDIT score of 8 or more

Exclusion Criteria:

* none

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 804 (Actual)
Dates: Start 2012-05; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Drinks in a typical week | 3 months
  Number of drinks in a typical week
AUDIT-C score | 3 months
  Composite measure of three drinking items - frequency of drinking, drinks per drinking day, frequency of 5+ drinking days
Highest number of drinks on one occasion | 3 months
  Highest number of drinks on one occasion in the past 3 months

CONTACTS AND LOCATIONS:
Overall Officials: John Cunningham, Ph.D., Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Cunningham JA, Murphy M, Hendershot CS. Treatment dismantling pilot study to identify the active ingredients in personalized feedback interventions for hazardous alcohol use: randomized controlled trial. Addict Sci Clin Pract. 2014 Dec 10;10(1):1. doi: 10.1186/s13722-014-0022-1. PMID 25539597
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching — http://www.camh.net/research